CLINICAL TRIAL: NCT02419118
Title: "Monoclonal Antibodies for Treatment of Multiple Myeloma. Present Status and Aspects of Effector Mechanisms With Emphasis on the CD38 Antibody Daratumumab "
Brief Title: "Monoclonal Antibodies for Treatment of Multiple Myeloma. Emphasis on the CD38 Antibody Daratumumab "
Acronym: DARA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 181114
Record Dates: First submitted 2015-02-12; First posted 2015-04-17 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; monoclonal antibody; Daratumumab
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — daratumumab; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dara len dex (Experimental): Daratumumab in combination with lenalidomide and dexamethasone
  Interventions: Drug: Daratumumab; Drug: Lenalidomide; Drug: Dexamethasone
- Len dex (Active Comparator): Lenalidomide in combination with dexamethasone
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Daratumumab — Treatment of myeloma patients with Daratumumab
  Other Names: CD38 monoclonal antibody; HuMax CD38
  Arms: Dara len dex
Drug: Lenalidomide — Treatment of myeloma patients
Drug: Dexamethasone — Treatment of myeloma patients

SUMMARY:
Daratumumab is a new treatment for patients with myeloma. While many patients benefit from this treatment some do not and the mechanism(s) of failure are poorly understood. This study aims to clarify aspects of resistance to treatment with daratumumab in order to improve patient outcomes in the future.

DETAILED DESCRIPTION:
The effector mechanisms of daratumumab have been extensively studied in vitro, but the in vivo correlates and key determinants of success or failure when daratumumab is used alone or in combination with lenalidomide for treatment of patients with myeloma have not been clarified.

There is potentially a wide spectrum of factors that may influence the quality and duration of response following treatment with daratumumab. The integrity of the patient's immune system may be important. Prior lines of chemotherapy or the myeloma disease itself may impair humural (i.e. complement) or cellular (i.e. ADCC) effector mechanisms that are of importance for the response to daratumumab. Also intrinsic properties of the tumor cells or interactions between myeloma cells and the bone marrow microenvironment could make the myeloma cells refractory to daratumumab.

A better understanding of these variables may enable us to improve the quality and duration of daratumumab-induced responses and make daratumumab-based therapies more effective in the near future.

ELIGIBILITY:
Inclusion Criteria:

* Accepted for a clinical trial with Daratumumab for myeloma

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2015-10-01 (Actual)

PRIMARY OUTCOMES:
Response by IMWG criteria | 4 weeks
  Assessed by M-component in blood and urine samples

SECONDARY OUTCOMES:
T cell subset numbers | 4 weeks
  Measured in bood and bone marrow aspirates

CONTACTS AND LOCATIONS:
Overall Officials: Torben Plesner, MD, Principal Investigator — Vejle Hospital
Locations (1):
- Department of Hematology Vejle Hospital, Vejle, Denmark

REFERENCES:
- [Result] Franssen LE, van de Donk NW, Emmelot ME, Roeven MW, Schaap N, Dolstra H, Hobo W, Lokhorst HM, Mutis T. The impact of circulating suppressor cells in multiple myeloma patients on clinical outcome of DLIs. Bone Marrow Transplant. 2015 Jun;50(6):822-8. doi: 10.1038/bmt.2015.48. Epub 2015 Mar 23. PMID 25798669
- [Result] Overdijk MB, Verploegen S, Bogels M, van Egmond M, Lammerts van Bueren JJ, Mutis T, Groen RW, Breij E, Martens AC, Bleeker WK, Parren PW. Antibody-mediated phagocytosis contributes to the anti-tumor activity of the therapeutic antibody daratumumab in lymphoma and multiple myeloma. MAbs. 2015;7(2):311-21. doi: 10.1080/19420862.2015.1007813. PMID 25760767